CLINICAL TRIAL: NCT04159844
Title: Evaluation of the Stiffness and Pressure Applied on the Lower Leg by a New Compression Bandage on Healthy Subjects
Acronym: FUSION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratoires URGO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: F-19-06-BD001
Record Dates: First submitted 2019-10-24; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: 3 separate sets :
  * URGOBD001 SSI compared with the SSI of a short stretch bandage
  * URGOBD001 SSI associated with wading bandage compared with the SSI of a short stretch bandage
  * URGOBD001 SSI compared with the SSI of a multi component bandage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Short stretch bandage (Active Comparator): Application with 50% overlap in combinaison with wading
  Interventions: Device: URGOBD001
- Multi componant bandage (Active Comparator): Application with 50% overlap
  Interventions: Device: URGOBD001
- Short stretch bandage bis (Active Comparator): Application with 50% overlap in combinaison with wading
  Interventions: Device: URGOBD001 associated with wading

INTERVENTIONS:
Device: URGOBD001 — Application with 50% overlapping
  Arms: Multi componant bandage; Short stretch bandage
Device: URGOBD001 associated with wading — Application with 50% overlapping in association with wading
  Arms: Short stretch bandage bis

SUMMARY:
This study evaluates the stiffness and interface pressures of a new compression system URGOBD001 on healthy subjects, compares with a short stretch bandage and a multi component bandage.

DETAILED DESCRIPTION:
Compression therapy is widely used in the treatment of chronic venous leg ulcers (VLUs). The clinical performance of a compression system depends on the apply pressure and the stiffness.

The static stiffness index (SSI) is defined by the difference in interface pressure measured when the subject is standing (working pressure) and the interface pressure measured when the subject is in the lying position (resting pressure).

ELIGIBILITY:
Inclusion Criteria:

* Subject with a body mass index of less than 30 (BMI = kg / m²),
* Subject presenting a healthy skin on both legs without any sign of dermatological lesion,
* Subject presenting a venous doppler of the lower limbs without detectable anomaly
* Subject with a ankle brachial pressure index (ABPI) greater than 0.9 and less than 1.3 for each of the lower limbs,
* Subject accepting to wear a compressive system on both legs for a period of three days.

Exclusion Criteria:

* Subject with chronic venous insufficiency whose stage is greater than or equal to 2 (CEAP classification of chronic venous diseases)
* Subject with type I or II diabetes
* Subject with lipoedema and / or dismorphic leg
* Subject presenting ankle ankylosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2019-11-29 (Estimated); Study Completion 2019-11-29 (Estimated)

PRIMARY OUTCOMES:
SSI(Static Stiffness Index) ≥ 10 mmHg | Hour 48 after the application
  % of subject with a SSI≥ 10 mmHg

SECONDARY OUTCOMES:
SSI (Static Stiffness Index) | From Hour 0 (Baseline) to Hour 72 (end of study) after application
  Evolution over time
Interface pressure under the bandage | From Hour 0 (Baseline) to Hour 72 after application
  Evolution over time
Slippage of the bandage in cm | From Hour 0 (Baseline) to Hour 72 (end of study) after application
  Assessed by measuring with a tape at each time (i) the length (L) from the top of the bandage to the floor, Slippage (cm) = L(Time 0) - L (Time i)

CONTACTS AND LOCATIONS:
Overall Officials: Benigni JP, MD, Principal Investigator — Intertek France clinical studies
Locations (1):
- Intertek France Clinical studies, Paris, France